CLINICAL TRIAL: NCT05422872
Title: Exploring What Psychological Safety Competencies Are Being Acquired During the Training Period of Healthcare Students: A Delphi Study of Trainee Mentors
Brief Title: Delphi Study on Psychological Safety Competencies in Healthcare Training Curricula
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Miguel Hernández University of Elche (Unknown); European Cooperation in Science and Technology, COST (Unknown); RheinMain University of Applied Science (Unknown); University of Tartu (Other); Tartu Health Care College (Unknown); LAB University of Applied Sciences (Unknown); University of Haifa (Other); Vilnius university hospital Sanatros klinikos (Unknown); University of Malta (Other); Universidade Nova de Lisboa (Other); Clinical Hospital Centre Zagreb (Other); Pavol Jozef Safarik University (Other); University of Belgrade (Other)
Responsible Party: Principal Investigator, José Joaquín Mira Solves, Professor, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: CA19113
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Psychological Safety; Knowledge, Attitudes, Practice
Keywords: Psychological Safety; Healthcare students; Delphi study; Knowledge, attitudes, skills; Trainee mentors
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Croatia: Twenty to twenty-five professionals assigned to Croatian healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Estonia: Twenty to twenty-five professionals assigned to Estonian healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Finland: Twenty to twenty-five professionals assigned to Finnish healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Germany: Twenty to twenty-five professionals assigned to German healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Israel: Twenty to twenty-five professionals assigned to Israeli healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Lithuania: Twenty to twenty-five professionals assigned to Lithuanian healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Malta: Twenty to twenty-five professionals assigned to Maltese healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Portugal: Twenty to twenty-five professionals assigned to Portuguese healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Slovakia: Twenty to twenty-five professionals assigned to Slovakian healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Spain: Twenty to twenty-five professionals assigned to Spanish healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study
- Serbia: Twenty to twenty-five professionals assigned to Serbian healthcare institutions (inpatient and outpatient settings, and community, and social care centers) who are responsible for mentoring and supervising residents and students during their clinical internships in the fields of family medicine, obstetrics, midwifery, pharmacy, surgery, and department of medicine.
  Interventions: Other: Delphi study

INTERVENTIONS:
Other: Delphi study — A Delphi study will be conducted with several rounds up to expert consensus.

SUMMARY:
Psychological safety refers to the shared belief that a work team can face complex challenges when there is an environment of mutual respect and trust. Thus, healthcare professionals provide safer care when causes and ways to avoid clinical errors can be discussed and analyzed without fear of criticism or sanctions. A psychological safety climate can be a determinant of patient safety. In this way, this provides safer care when it is possible to discuss and analyze the causes and how to avoid clinical errors without fear of criticism or sanctions.

This study aims to explore the mentors' opinion on what psychological safety competencies are being acquired by future generations of healthcare professionals (students and residents, hereafter "trainees") through current training programs and what actions should be taken to promote such competencies in clinical settings.

DETAILED DESCRIPTION:
Consensus study based on the Delphi technique. To develop the questionnaire 0 structured interviews will be conducted. This study step includes the development of a consultation instrument in questionnaire format to conduct the Delphi study. Only the legibility, face and content validity of the questionnaire will be assessed through interviews to ensure its correct completion by the participants.

One member of the research team for each participating country will act as national study coordinator in that country.

The study procedure will be structured in the following steps:

1. Research team constitution.
2. Request for study evaluation and approval by an Ethics Committee in each of the participating countries. This step is required only in the case of countries where ethical evaluation is mandatory to conduct this type of study. A common draft of the protocol will be available to support each national coordinator.
3. Collect preliminary information for the subsequent questionnaire re-define for the Delphi study. For this purpose, the available literature on the topic of the study and the WHO Global Patient Safety Action Plan 2021-2030 (more specifically, objective 5) has been reviewed beforehand. Once the first version of the questionnaire has been drafted from the information collected, interviews will be conducted with 3 mentors from each participating country to assess the legibility, face, and content validity of the draft questionnaire (readability, comprehension, clarity, coherence, relevance, and appropriateness). A template will be available to conduct it.
4. Revision and improvement of the initial version of the questionnaire based on the information gathered through the interviews to ensure the face and content validity of the instrument.
5. Approval of the questionnaire by the research team based on the information collected in steps 3 and 4. The questionnaire will be translated from English into the local languages of the participating countries by two native experts independently. Inconsistencies will be resolved with the participation of a third researcher.
6. Recruitment of participants. The national coordinator will be responsible for contacting the teaching units of healthcare institutions in their country to establish, through them, contact with trainees' mentors. A minimum of 20 participants from each country is expected. They will be working in family medicine, midwifery, pharmacy, surgery, and medicine departments.
7. Invitation to the study. The questionnaire will be designed on a web platform, property of the research team, hosted on a secure server, and specifically designed for conducting Delphi studies. The responses given to the questionnaire will be treated as fully confidential. However, given the nature of the study (Delphi with several rounds), each participant will access the web platform through personalized credentials to allow continuity in data collection and analysis. Personal information (username and password) will be deleted, and the responses of the same person to the different rounds will be linked by a unique double-blind code. The questionnaire will be disseminated by e-mail. Three reminders are foreseen to ensure an adequate response rate.
8. First round and successive rounds up to expert consensus. A minimum of two rounds will be carried out, and the maximum will be determined by reaching a consensus among the participants.
9. Data analysis and interpretation of the results. Preparation of an article for publication in a scientific journal.
10. Dissemination of the results. The results will be translated into practice to improve the training programs of next generations of health professionals through schools and faculties, ministries of health, and other agencies and scientific societies involved in curricula design. The results will also be disseminated through the usual scientific media (journals, conferences, etc.) and social networks.

ELIGIBILITY:
Inclusion Criteria:

* Trainees mentors in healthcare institutions (inpatient and outpatient settings, and community and social care centers) in Croatia, Estonia, Finland, Germany, Israel, Lithuania, Malta, Portugal, Serbia, Slovakia, and Spain.
* Working in inpatient or outpatient settings or community or social care centers mentoring residents in the fields of family medicine, midwifery, pharmacy, surgery, and medicine department.

Exclusion criteria:

• Academic mentors. The study setting is social and health care centers, not academia.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Trainees' mentors who would be working in inpatient or outpatient settings or community or social care centers mentoring residents in the fields of family medicine, midwifery, pharmacy, surgery, and medicine department.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Psychological safety competencies - Degree of KNOWLEDGE acquisition (round 1) | Data collection for the first round of the Delphi study will extend from the start of the study for 20 days.
  What knowledge in psychological safety is being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 7 items referring to knowledge. Participants (mentors of healthcare trainees) will have to assess each knowledge (competence component) according to its degree of acquisition (5-point Likert scale).
Psychological safety competencies - Degree of significance of KNOWLEDGE (round 1) | Data collection for the first round of the Delphi study will extend from the start of the study for 20 days.
  What knowledge in psychological safety is being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 7 items referring to knowledge. Participants (mentors of healthcare trainees) will have to assess each knowledge (competence component) according to its degree of significance (5-point Likert scale).
Psychological safety competencies - Degree of ATTITUDE acquisition (round 1) | Data collection for the first round of the Delphi study will extend from the start of the study for 20 days.
  What attitudes toward psychological safety are being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 6 items referring to attitudes. Participants (mentors of healthcare trainees) will have to assess each attitude (competence component) according to its degree of acquisition (5-point Likert scale).
Psychological safety competencies - Degree of significance of the ATTITUDE (round 1) | Data collection for the first round of the Delphi study will extend from the start of the study for 20 days.
  What attitudes toward psychological safety are being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 6 items referring to attitudes. Participants (mentors of healthcare trainees) will have to assess each attitude (competence component) according to its degree of significance (5-point Likert scale).
Psychological safety competencies - Degree of SKILL acquisition (round 1) | Data collection for the first round of the Delphi study will extend from the start of the study for 20 days.
  What psychological safety skills are being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 7 items referring to skills. Participants (mentors of healthcare trainees) will have to assess each skill (competence component) according to its degree of acquisition (5-point Likert scale).
Psychological safety competencies - Degree of significance of the SKILL (round 1) | Data collection for the first round of the Delphi study will extend from the start of the study for 20 days.
  What psychological safety skills are being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 7 items referring to skills. Participants (mentors of healthcare trainees) will have to assess each skill (competence component) according to its degree of significance (5-point Likert scale).
Psychological safety INTERVENTIONS - Degree of implementation (round 1) | Data collection for the first round of the Delphi study will extend from the start of the study for 20 days.
  What actions the healthcare institutions in which the trainees do their clinical internships should implement to promote the acquisition of these competencies.
  Participants (mentors of healthcare trainees) will have to assess each intervention according to its degree of implementation in their center (5-point Likert scale).
Psychological safety INTERVENTIONS - Degree of significance (round 1) | Data collection for the first round of the Delphi study will extend from the start of the study for 20 days.
  What actions the healthcare institutions in which the trainees do their clinical internships should implement to promote the acquisition of these competencies.
  Participants (mentors of healthcare trainees) will have to assess each intervention according to its degree of significance (5-point Likert scale).
Psychological safety competencies - Degree of KNOWLEDGE acquisition (round 2) | Twenty-seven days after initiating the study, the second round of the Delphi study will extend for 20 days.
  What knowledge in psychological safety is being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 7 items referring to knowledge. Participants (mentors of healthcare trainees) will have to assess each knowledge (competence component) according to its degree of acquisition (5-point Likert scale).
Psychological safety competencies - Degree of significance of KNOWLEDGE (round 2) | Twenty-seven days after initiating the study, the second round of the Delphi study will extend for 20 days.
  What knowledge in psychological safety is being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 7 items referring to knowledge. Participants (mentors of healthcare trainees) will have to assess each knowledge (competence component) according to its degree of significance (5-point Likert scale).
Psychological safety competencies - Degree of ATTITUDE acquisition (round 2) | Twenty-seven days after initiating the study, the second round of the Delphi study will extend for 20 days.
  What attitudes toward psychological safety are being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 6 items referring to attitudes. Participants (mentors of healthcare trainees) will have to assess each attitude (competence component) according to its degree of acquisition (5-point Likert scale).
Psychological safety competencies - Degree of significance of the ATTITUDE (round 2) | Twenty-seven days after initiating the study, the second round of the Delphi study will extend for 20 days.
  What attitudes toward psychological safety are being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 6 items referring to attitudes. Participants (mentors of healthcare trainees) will have to assess each attitude (competence component) according to its degree of significance (5-point Likert scale).
Psychological safety competencies - Degree of SKILL acquisition (round 2) | Twenty-seven days after initiating the study, the second round of the Delphi study will extend for 20 days.
  What psychological safety skills are being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 7 items referring to skills. Participants (mentors of healthcare trainees) will have to assess each skill (competence component) according to its degree of acquisition (5-point Likert scale).
Psychological safety competencies - Degree of significance of the SKILL (round 2) | Twenty-seven days after initiating the study, the second round of the Delphi study will extend for 20 days.
  What psychological safety skills are being acquired by future generations of healthcare professionals (students and residents referred to as "trainees") through their clinical internships.
  The questionnaire contains 7 items referring to skills. Participants (mentors of healthcare trainees) will have to assess each skill (competence component) according to its degree of significance (5-point Likert scale).
Psychological safety INTERVENTIONS - Degree of implementation (round 2) | Twenty-seven days after initiating the study, the second round of the Delphi study will extend for 20 days.
  What actions the healthcare institutions in which the trainees do their clinical internships should implement to promote the acquisition of these competencies.
  Participants (mentors of healthcare trainees) will have to assess each intervention according to its degree of implementation in their center (5-point Likert scale).
Psychological safety INTERVENTIONS - Degree of significance (round 2) | Twenty-seven days after initiating the study, the second round of the Delphi study will extend for 20 days.
  What actions the healthcare institutions in which the trainees do their clinical internships should implement to promote the acquisition of these competencies.
  Participants (mentors of healthcare trainees) will have to assess each intervention according to its degree of significance (5-point Likert scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo ATENEA, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
The databases, without identification and code registration, will be available at OSF (Center for Open Science) for access by the scientific community. the scientific community.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Six months after the data collecting.
Access Criteria: Data repository is available for the scientific community.

REFERENCES:
- [Background] O'Donovan R, McAuliffe E. A systematic review exploring the content and outcomes of interventions to improve psychological safety, speaking up and voice behaviour. BMC Health Serv Res. 2020 Feb 10;20(1):101. doi: 10.1186/s12913-020-4931-2. PMID 32041595
- [Background] Richard A, Pfeiffer Y, Schwappach DDL. Development and Psychometric Evaluation of the Speaking Up About Patient Safety Questionnaire. J Patient Saf. 2021 Oct 1;17(7):e599-e606. doi: 10.1097/PTS.0000000000000415. PMID 28858000
- [Background] Schwappach D, Sendlhofer G, Hasler L, Gombotz V, Leitgeb K, Hoffmann M, Jantscher L, Brunner G. Speaking up behaviors and safety climate in an Austrian university hospital. Int J Qual Health Care. 2018 Nov 1;30(9):701-707. doi: 10.1093/intqhc/mzy089. PMID 29701770
- [Background] Schwappach D, Sendlhofer G, Kamolz LP, Kole W, Brunner G. Speaking up culture of medical students within an academic teaching hospital: Need of faculty working in patient safety. PLoS One. 2019 Sep 12;14(9):e0222461. doi: 10.1371/journal.pone.0222461. eCollection 2019. PMID 31514203
- [Background] Derickson R, Fishman J, Osatuke K, Teclaw R, Ramsel D. Psychological safety and error reporting within Veterans Health Administration hospitals. J Patient Saf. 2015 Mar;11(1):60-6. doi: 10.1097/PTS.0000000000000082. PMID 24583957
- See also: COST (European Cooperation in Science and Technology) — http://www.cost.eu